CLINICAL TRIAL: NCT01605110
Title: Effects of HBOT for Edema/Ecchymosis After Upper Eyelid Blepharoplasty (Single Site Study)
Brief Title: Effects of Hyperbaric Oxygen Therapy on Surgical Wound Healing
Acronym: BLEPH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Restorix Research Institute, LLLP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RRI-2011-02-BLEPH-00 BS
Record Dates: First submitted 2011-09-02; First posted 2012-05-24 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Edema; Ecchymosis
Keywords: blepharoplasty; hyperbaric; oxygen; ecchymosis; edema; wound; healing
MeSH Terms: conditions — Edema; Ecchymosis; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperbaric oxygen therapy (Experimental): We propose to study the effects of two HBOT treatments (one before and one after surgery) with patients who have undergone upper eyelid surgery. Reduction in swelling and bruising will be assessed at 3, 10, 21, 30 and 90 days post-surgery to determine if healing is accelerated by HBOT. Patients that volunteer to participate in this study will be exposed to two treatments of 100% oxygen at 2.0 atmospheres absolute (ATA) or air (sham) 1.2 ATA inside mono-place chambers for 90 minutes. By comparing oxygen treatment groups with a matched control group, we can accurately assess the effectiveness of this treatment for patients. By participating in this study, patients will help in establishing the best treatment practices of using HBOT to accelerate healing and reduce cost in surgical recovery.
  Interventions: Drug: Hyperbaric oxygen treatment
- Air sham (Sham Comparator): We propose to study the effects of two HBOT treatments (one before and one after surgery) with patients who have undergone upper eyelid surgery. Reduction in swelling and bruising will be assessed at 3, 10, 21, 30 and 90 days post-surgery to determine if healing is accelerated by HBOT. Patients that volunteer to participate in this study will be exposed to two treatments of 100% oxygen at 2.0 atmospheres absolute (ATA) or air (sham) 1.2 ATA inside mono-place chambers for 90 minutes. By comparing oxygen treatment groups with a matched control group, we can accurately assess the effectiveness of this treatment for patients. By participating in this study, patients will help in establishing the best treatment practices of using HBOT to accelerate healing and reduce cost in surgical recovery.
  Interventions: Drug: Air sham

INTERVENTIONS:
Drug: Hyperbaric oxygen treatment — Patients that volunteer to participate in this study will be exposed to two treatments (one before surgery; one after surgery) of 100% oxygen at 2.0 atmospheres absolute (ATA) inside mono-place chambers for 90 minutes (at depth).
  Arms: Hyperbaric oxygen therapy
Drug: Air sham — Patients that volunteer to participate in this study will be exposed to two treatments (one before surgery; one after surgery) of medical grade air (21%oxygen; sham) at 1.2 ATA inside mono-place chambers for 90 minutes.
  Arms: Air sham

SUMMARY:
The aim of this study is to test the effect of Hyperbaric Oxygen Therapy) HBOT (100% oxygen; 2.0 ATA; 90 minute total exposure) and compare against a hyperbaric sham treatment (HBST) (patient's breathing room air; 2.0 ATA; 90 minute exposure) in reducing edema and ecchymosis. HBOT will be applied as a single pre-operative and a single post-operative treatment for patients undergoing eyelid surgery. Briefly, patients will be exposed to HBOT 2-4 hours prior to undergoing surgery, 2-4 hours post-surgery and healing will be assessed at day 3, 10, 21, 30 & 90 days after surgery. Edema and ecchymosis will be assessed in a time series to determine the extent that HBOT reduces these clinical signs. The primary null hypothesis to test will be that no differences in scores will exist between treatment and control at day 3, 10 & 21 post-surgery. A secondary null hypothesis to test is the time required to change a score will be no different between the two groups.

HBOT=hyperbaric oxygen therapy; HBST=hyperbaric sham treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients that are able to undergo surgery at the Allure Clinic are capable of undergoing exposure to HBOT, as the contraindications of HBOT are similar to eyelid surgery, with few exceptions.

Exclusion Criteria:

* The investigators will exclude active smokers and those who have quit smoking in the last 12 months, those with known lung disease, seizure disorder, congestive heart failure, known active cancer, previous treatment with specific chemotherapy agents (Doxorubicin, Bleomycin, Disulfiram, Cis-platinum, Mafenide acetate), those who cannot undergo pressurization/ depressurization because of eustachian-tube dysfunction and confinement anxiety.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
A measureable reduction of ecchymosis grade in treatment group vs. control group | 21 days
  Ecchymosis will be assessed in a time series to determine the extent that HBOT reduces these clinical signs. The primary null hypothesis to test will be that no differences in scores will exist between treatment and control at day 3, 10 & 21 post-surgery.

SECONDARY OUTCOMES:
A measureable reduction of edema grade in treatment group vs. control group | 21 days
  Edema will be assessed in a time series to determine the extent that HBOT reduces these clinical signs. The primary null hypothesis to test will be that no differences in scores will exist between treatment and control at day 3, 10 & 21 post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Sires, MD, FACS, Principal Investigator — Allure Laser Center & Medispa
Locations (1):
- Restorix Research Institute, Issaquah, Washington, United States